CLINICAL TRIAL: NCT00174694
Title: A Prospective, Randomized, Open-label, Active-controlled Study in Adult Subjects With Acute Bacterial Sinusitis Comparing the Clinical Efficacy of Telithromycin (KETEK®) 800 mg Once a Day for 5 Days Versus Amoxicillin-clavulanic Acid (AUGMENTIN®) 875/125 mg Twice a Day for 10 Days
Brief Title: CHOOSE : Telithromycin, Acute Bacterial Sinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR3647A_4023; EudraCT # : 2004-001460-42
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — telithromycin

INTERVENTIONS:
Drug: Telithromycin

SUMMARY:
Primary objective:

* To demonstrate that the clinical efficacy of telithromycin (800 mg od for 5 days) is non-inferior to amoxicillin-clavulanic acid (875/125 mg bid for 10 days) at the test-of-cure (TOC) visit (Day 17-21) in subjects with acute bacterial sinusitis (ABS).

Secondary objective(s):

* To assess the time to resolution of signs and symptoms between the baseline (Day 1) and TOC (Day 17-21) visits,
* To assess the rate of clinical relapse at the follow-up visit (Day 41-49),
* To assess health economic outcome until follow-up visit (Day 41-49),
* To assess quality of life up to the follow-up visit (Day 41-49),
* To compare the safety of telithromycin and amoxicillin-clavulanic acid,
* To compare the bacteriologic outcome of both treatments as observed at TOC (Day 17-21) and at follow-up visit (Day 41-49),in subjects with ABS.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant female
* Outpatients with a clinical diagnosis of ABS, based on the presence of:

  * Signs and symptoms lasting longer than 7 days and less than 28 days,
  * Purulent anterior or posterior nasal discharge
  * One additional major sign and symptom or 2 minor signs and symptoms. The major and minor signs and symptoms will be defined as the following:

    * Major signs and symptoms: facial pain/pressure/tightness over the maxillary sinuses, nasal congestion/obstruction, change in the perception of smell (hypoanosmia/anosmia), fever (temperature > 38° C [100.4 F] (oral)/ > 38.5° C [101.2 F] (tympanic)/ > 39° C [102.2 F] (rectal)),
    * Minor signs and symptoms: headache, halitosis, dental pain, ear pressure/fullness, cough, fatigue,
* Subjects with abnormal maxillary sinus x-rays (Waters views and additional views if necessary) or limited sinus CT scans or sinus ultrasound in the previous 48 hours before inclusion defined as the presence of at least 1 of the following homolateral radiological criteria:

  * Presence of air/fluid level,
  * Total opacification,
  * Mucosal thickening > 10 mm, Written informed consent must be obtained before enrollment in the study for all subjects.

Exclusion Criteria:

* Related to the disease :

  * History of recurrent sinusitis (more than (>) 3 episodes of sinusitis requiring antibiotic therapy within the previous 12 months),
  * Chronic sinusitis (signs and symptoms lasting more than 28 days),
  * Suspicion of sinusitis requiring treatment other than oral antibiotic therapy,
  * Suspicion of concomitant odontologic infection, requiring antibiotic therapy or surgery
  * Nosocomial sinusitis (eg, hospitalization more than 48 hours or non ambulatory institutional confinement including nursing homes within 2 weeks),
  * Known major obstructive anatomic/functional lesions in nasopharynx: anatomical blockage (eg, chronic nasal polyps, severely deviated septum), cystic fibrosis, immotile cilia, sinus polyps,
  * Use of nasal, nasogastric or nasotracheal catheters,
  * Sinus puncture and/or sinus lavage in the previous 7 days,
  * Previous sinus surgery in the last 6 months,
  * Maxillary sinusitis requiring immediate surgery
  * Symptomatic allergic sinusitis and/or allergic rhinitis,
  * Exposition to environmental irritants in the workplace
* Related to the previous/concomitant medication :

  * Previous treatment with intranasal, oral or parenteral antibiotic (more than 24 hours intake) within 30 days prior enrollment,
  * Intranasal corticosteroid or short term systemic corticosteroid use within the past 10 days prior to enrollment,
  * Maintenance systemic corticosteroid therapy on inclusion (>10 mg/day equivalent prednisone),
  * Subjects who are long-term users (> 4 weeks) of nasal decongestants like oxymetazoline 0.05%,
  * Required on-therapy contra-indicated medications with study treatment (according to the country labeling): ergot alkaloids derivatives (such as ergotamine and dihydroergotamine), cisapride, pimozide, astemizole, terfenadine, simvastatin, atorvastatin and lovastatin, allopurinol, methotrexate, probenecid,
  * Previous treatment within 2 weeks before enrollment or during the study medication with rifampicin, phenytoin, carbamazepine, St-John's-wort, phenobarbital,
  * Treatment with any investigational product in the last 30 days before study entry.
* Other exclusion criteria

  * Subject with mononucleosis, phenylketonuria,
  * Immunocompromised subjects, such as: subjects with known HIV subjects and those who have either had an AIDS-defining condition (eg, Kaposi's sarcoma, Pneumocystis carinii pneumonia) or have CD4+ T-lymphocyte count < 200/mm3, known neutropenia (< 1500 neutrophils/mm3) not attributable to the acute infectious disease, metastatic or hematological malignancy, splenectomized or known hyposplenia or asplenia,
  * History of congenital or a family history of long QT syndrome (if not excluded by previous ECG),
  * Subjects with known acquired QT interval prolongation,
  * Subjects with myasthenia gravis,
  * Subjects with galactose intolerance,
  * Subjects with a progressively fatal disease, life expectancy £ 3 months,
  * Women who are breast-feeding or are pregnant or childbearing potential (ie, ovulating, premenopausal, not surgically sterile) or who are failing to use adequate contraception for example systemic hormones (birth control pills, implant), intrauterine device or barrier method (diaphragm with intravaginal spermicide, cervical cap, male or female condom). A urine or serum test will be carry out before enrollment in the study,
  * History or known hypersensitivity and/or adverse reactions to telithromycin or macrolides, amoxycillin-clavulanic acid or betalactams,
  * Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult,
  * History of drug or alcohol abuse rendering subjects unable to comply with protocol,
  * Known or history of severe impaired renal function, as shown by a previous laboratory value of creatinine clearance ≤ 30 ml/min either measured or estimated with Cockroft formula or serum creatinine > or =2.0 mg/dL (> or =176 μmol/L),
  * Mental condition rendering the subjects unable to understand the nature, scope, and possible consequences of the study,
  * Subjects unlikely to adhere to the protocol, eg, uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study,
  * Subject is the investigator or any subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof involved in the conduct of the protocol,
  * Subjects having already been included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2004-11; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
clinical success rate at the TOC visit in the per protocol population. | During all the study conduct

SECONDARY OUTCOMES:
Time of regression of signs and symptoms of sinusitis, rate of clinical relapse at follow-up visit.Bacteriological data.Safety data... | During all the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Perdriset, MD, Study Director — Sanofi

REFERENCES:
- [Result] Desrosiers M, Ferguson B, Klossek JM, Drugeon H, Mosges R. Clinical efficacy and time to symptom resolution of 5-day telithromycin versus 10-day amoxicillin-clavulanate in the treatment of acute bacterial sinusitis. Curr Med Res Opin. 2008 Jun;24(6):1691-702. doi: 10.1185/03007990802133914. PMID 18559163